CLINICAL TRIAL: NCT04793230
Title: Predictive Value of Nasolacrimal Sac Biopsy in Endoscopic Dacryocystorhinostomy
Brief Title: Nasolacrimal Sac Biopsy in Endoscopic Dacryocystorhinostomy
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abdulkarim Hasan, pathology laboratory coordinator, Al-Azhar University
Other Study IDs: 19-11-002
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Dacryocystitis; Chronic
MeSH Terms: conditions — Dacryocystitis; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: biopsying — The procedure was carried out under general or local anesthesia. An otolaryngologist conducts the endoscopic intranasal operation, while an eye surgeon removes tissue from the sac and lacrimal tubes using lacrimal probes passed through the canaliculi.

SUMMARY:
During dacryocystorhinostomy (DCR), the lacrimal sac wall biopsy is not routinely performed, but it is recommended if there is a suspicion of underlying disease other than preoperatively or intraoperatively chronic inflammation. We aimed to evaluate the utility of the histopathology examination of fifty patients in AlAzhar Hospitals to put recommendation for histopathology examination of such cases.

DETAILED DESCRIPTION:
Most of patient with epiphora have different causes of nasolacrimal duct obstruction . This study aims to examine how important routine lacrimal sac biopsy is during endoscopic dacryocystorhinostomy surgery.

The study included 50 patients with chronic unilateral epiphora. All patients underwent endoscopic dacryocystorhinostomy with nasolacrimal duct biopsy. Histopathologic analysis was performed for each specimen to assess the nature of the pathology.

ELIGIBILITY:
Inclusion Criteria:

- Male and female patients with chronic lacrimal duct obstruction attended the outpatient clinic of the hospital for treatment during the study period.

Exclusion Criteria:

* Patients refusing the biopsy
* Patients asked for histopathology in private laboratories

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes fifty patients with chronic epiphora due to chronic nasal duct obstruction seeking for treatment by endoscopic intranasal dacryocystorhinostomy. Their age ranged from (20-70) years from both genders. They were selected from patients attending the Ophthalmology and Ear Nose Throat (ENT) clinics, at Al-Azhar University Hospital. Their referring ophthalmologist diagnosed all of the patients with lacrimal obstruction.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-03-09 (Actual)

PRIMARY OUTCOMES:
Microscopic examination using Hematoxylin and Eosin stains with special stain | fourteen days
  sending the biopsies to the pathology laboratory with completed request form then examination of the biopsies in the laboratory using the light microscope to assess the nature of the lesion with degree of inflammation according to the amount of lymphocytes to be classified as mild (10% cells), moderate (up to 50%) or severe (more than 50% lymphocytic cells)

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim El-dsoky, MD, Principal Investigator — Al-Azhar University
Locations (1):
- Azhar faculty of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
journal pubication